CLINICAL TRIAL: NCT02752087
Title: A Study to Compare the Pharmacokinetics and Pharmacodynamics of LY900014 Test Versus Reference Formulations in Healthy Subjects
Brief Title: A Study to Compare the Effects of a Test and Reference Formulation of LY900014 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16489; I8B-MC-ITRP (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2016-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- U-193 LY900014 Test (Experimental): LY900014 test dose administered via subcutaneous (SC) injection
  Interventions: Drug: LY900014
- U-95 LY900014 Reference (Active Comparator): LY900014 reference dose administered via SC injection
  Interventions: Drug: LY900014

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro

SUMMARY:
This study of healthy participants evaluated the concentration of a test LY900014 and a reference LY900014 formulation in the bloodstream and how it affected the blood sugar levels. The whole study, including screening, took up to 8 weeks to complete.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who can potentially get pregnant:

  * Must have a negative pregnancy test at the time of screening
  * Agree to continue to use a reliable method of birth control until the end of the study
* Have a body mass index (BMI) of 18.0 to 30.0 kilogram per meter square (kg/m²), inclusive, at screening
* Are nonsmokers, have not smoked for at least 2 months before entering the study

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to insulin lispro, related compounds, or any components of the formulation
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Intend to use over-the-counter or prescription medication within 7 and 14 days, respectively, before dosing (apart from vitamin/mineral supplements, occasional paracetamol, hormonal contraception, or thyroid-replacement therapy)
* Have used systemic glucocorticoids within 3 months prior to entry into the study
* Have donated blood of more than 450 milliliters (mL) or more in the last 3 months or provided any blood donation within the last month before screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a four-period crossover study of U-193 LY900014 test formulation and U-95 LY900014 reference formulation with a minimum of 3 days between dosing.
Groups:
- LY900014 Test/Reference/Test/Reference: U-193 LY900014 test formulation administered once subcutaneously (SC) in Study Periods 1 and 3. U-95 LY900014 reference formulation administered once SC in Study Periods 2 and 4.
- LY900014 Reference/Test/Reference/Test: U-95 LY900014 reference formulation administered once SC in study periods 1 and 3. U-193 LY900014 test formulation administered once SC in study periods 2 and 4.
Period: Study Period 1
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 12 | 12
Received Study Drug | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Study Period 2
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 11 | 12
Received Study Drug | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Washout
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Study Period 3
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 11 | 12
Received Study Drug | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Washout
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Study Period 4
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 11 | 12
Received Study Drug | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | LY900014 Test/Reference/Test/Reference | LY900014 Reference/Test/Reference/Test
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: U-193 LY900014 test formulation administered once SC in 2 of 4 study periods. U-95 LY900014 reference formulation administered once SC in 2 of 4 study periods.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 8 Hours (AUC[0-8 Hours])
Description: PK: Insulin Lispro Area Under the Concentration Curve From Time Zero to 8 Hours (AUC[0-8 Hours])
Time Frame: 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, 360, 420, and 480 minutes post study dose for each treatment
Population: All participants who completed at least 1 study period and had measurable insulin lispro concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour/liter (pmol*h/L)
Units Other Than Participants: Number of observations
Groups:
- LY900014 Reference: U-95 LY900014 reference formulation administered once SC in 2 of 4 study periods.
- LY900014 Test: U-193 LY900014 test formulation administered once SC in 2 of 4 study periods.
Arm/Group | LY900014 Reference | LY900014 Test
Number analyzed (Participants) | 23 | 24
Number analyzed (Number of observations) | 46 | 47
picomole*hour/liter (pmol*h/L) | 2440 (13) | 2430 (13)

2. Secondary Outcome: Pharmacodynamics (PD): Total Amount of Glucose Infused (Gtot)
Description: Gtot is the total glucose infusion over the clamp duration. It is used to measure the study drug action over time as measured by the euglycemic clamp procedure.
Time Frame: Blood glucose was measured approximately every 2.5 minutes for the first 30 minutes, then every 5 minutes until 120 minutes post dose, and then every 10 minutes until 480 minutes post dose
Population: All participants who completed at least 1 clamp procedure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram (mg)
Units Other Than Participants: Number of observations
Arm/Group | LY900014 Reference | LY900014 Test
Number analyzed (Participants) | 23 | 24
Number analyzed (Number of observations) | 46 | 47
milligram (mg) | 108,000 (34) | 117,000 (35)

ADVERSE EVENTS:
Arm/Group | LY900014 Test | LY900014 Reference
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 9/24 | 8/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 Test (N=24) | LY900014 Reference (N=23)
Infusion site erythema (General disorders) | 2 (2) | 0 (0)
Infusion site swelling (General disorders) | 3 (5) | 3 (3)
Injection site erythema (General disorders) | 1 (1) | 2 (3)
Injection site pain (General disorders) | 2 (2) | 3 (3)
Vessel puncture site bruise (General disorders) | 5 (9) | 1 (1)
Vessel puncture site rash (General disorders) | 2 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes